CLINICAL TRIAL: NCT06649123
Title: Development of a Multiomics Assay for Use on OriColTM Sampled Rectal Mucus for Detection of Cancer and Significant Polyps in Symptomatic Patients on the Colorectal Urgent Suspected Cancer Pathway
Brief Title: Triple Assay of Rectal Mucus in the Diagnosis of Colorectal Cancer
Acronym: TRIOMIC
Status: Recruiting | Type: Observational
Sponsor: Origin Sciences (Industry)
Collaborators: Shrewsbury and Telford Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: Oricol-EGI-04
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer; Adenoma Colon Polyp
Keywords: colon; rectum; mucus; adenoma; microbiome
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sample of rectal mucus containing shed cells from the gastrointestinal tract, microbiome and breakdown products of digestion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Oricol Test — Assessment of diagnostic accuracy of Oricol Sampling device for triage in patients with suspected lower gastrointestinal cancer

SUMMARY:
Development of a multiomics assay for use on OriColTM sampled rectal mucus for detection of cancer and significant polyps in symptomatic patients on the Colorectal Urgent Suspected Cancer pathway.

DETAILED DESCRIPTION:
The primary objectives of the study are:

1. Confirm the presence of established genetic, epigenetic and microbiome based biomarker signatures associated with CRC and high-risk adenoma (defined as >10mm in diameter or the presence of high-grade dysplasia) in colorectal urgent suspected cancer referrals, who are triaged for colonoscopy.
2. To expand and refine the genomic, epigenetic and microbiome biomarker signature profiles associated with colorectal cancer and high-risk adenoma to identify rarer biomarkers in addition to those previously established.
3. To generate indicative performance metrics, including an assessment of discriminatory power, sensitivity, specificity and negative predictive values for the clinical application of Oricol™ multiomics assay.

The Secondary Objectives of the study are:

1. To assess the health economics of delivering a diagnostic service to patients referred to the urgent suspected cancer (USC) pathway via a Community Diagnostic Centre (CDC) in comparison to the current delivery mechanisms through the Two-Week Wait (TWW) pathway.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years and over
2. Patients referred from primary care to the 'urgent suspected cancer' CRC pathway during the study period.
3. Patients who provide voluntary written informed consent to participate in the study.

Exclusion Criteria:

1. Patients who are unable to undergo digital rectal examination (DRE).
2. Patients with peri-anal/anal symptoms that may limit DRE and proctoscopy examination and it would be clinically inappropriate to attempt to assess these patients. This may include conditions such as:

   * Patients who have undergone radiotherapy.
   * An acute or chronic anal fissure
   * Perianal haematoma
   * Acute thrombosed haemorrhoids
   * Post- operative anal stenosis
   * The presence of an obstructing anal/low rectal tumour or discomfort as a result of previous pelvic radiotherapy
3. Current pregnancy or suspicion of pregnancy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 6600 patients referred through the UK Urgent Suspected Cancer Pathway.
Sampling Method: Non-Probability Sample
Enrollment: 6600 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
TRIOMIC - 1 | 26 months
  Determination of the clinical utility for stratification of colorectal cancer and high risk adenoma in a symptomatic population using hologenomic analysis.
TRIOMIC - 2 | 26 month
  To expand and refine the genomic, epigenetic and microbiome biomarker signature profiles associated with colorectal cancer and high-risk adenoma to identify rarer biomarkers in addition to those previously established.
TRIOMIC - 3 | 26 months
  To generate indicative performance metrics, including an assessment of discriminatory power, sensitivity, specificity and negative predictive values for the clinical application of Oricol™ multiomics assay.

SECONDARY OUTCOMES:
Health Economic Assessment | 26 months
  1. To assess the health economics of delivering a diagnostic service to patients referred to the urgent suspected cancer (USC) pathway via a Community Diagnostic Centre (CDC) in comparison to the current delivery mechanisms through the Two-Week Wait (TWW) pathway.

CONTACTS AND LOCATIONS:
Locations (1):
- Shrewsbury & Telford NHS Foundation Trust, Telford, Shropshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
As this study is supporting development of assay for diagnostics, the data will not be shared until completion of the research.

REFERENCES:
- [Background] Humphrey HN, Diodato A, Isner JC, Walker E, Lacy-Colson J, Nedjai B, Daniels IR; ORI-EGI-02 Study Group. An internal pilot study of a novel rectal mucocellular sampling device to allow next-generation sequencing for colorectal disease. Tech Coloproctol. 2023 Mar;27(3):227-235. doi: 10.1007/s10151-022-02704-y. Epub 2022 Sep 27. PMID 36166177